CLINICAL TRIAL: NCT06577129
Title: Effects of Ladder Training Versus Plyometric Training Program on Agility, Speed and Power in Domestic Female Cricket Players
Brief Title: Effects of Ladder Training Versus Plyometric Training Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: F22C14G79010
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Sports Physical Therapy
Keywords: Ladder training, plyometric, female domestic players
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ladder training (Experimental): Participants 21 out of 42 received ladder training.
  Interventions: Other: Ladder training
- Plyometric training (Active Comparator): 21 participants out of 42 received ladder training.
  Interventions: Other: Plyometric training

INTERVENTIONS:
Other: Ladder training — Players exercised three times a week for sixty minutes apiece on a ladder for eight weeks. The drills were divided into three categories: steady state drills, burst drills, and elastic reaction drills. While steady state training focused on agility and endurance, burst drills were more focused on fast foot movement. Elastic response drills targeted the reactive speed components of the lower leg.
  Arms: Ladder training
Other: Plyometric training — For eight weeks, the players performed a 60-minute plyometric training program three times a week. A fifteen-minute warm-up, stretching, and jogging session comes after the thirty minutes of plyometric training. The cool-down consists of fifteen minutes of light running and stretching.
  Arms: Plyometric training

SUMMARY:
A team sport such as cricket consists of irregular sequences of high- and low-intensity motions utilising different metabolic pathways. Athlete performance in this sport is correlated with every facet of physical fitness, including muscular strength, agility, speed, anaerobic power (vertical leap), and aerobic capacity. All aspects of physical fitness, such as aerobic capacity, anaerobic power (vertical leap), agility, speed, and muscular strength, are related to success in this sport. Plyometric training that is repetitive and intermittent has been recommended as a useful tactic for cricket-specific training regimens. Plyometric exercise training is a type of workout regimen designed to enhance nervous system functioning and generate powerful, quick movements, ultimately improving sports performance. Plyometric training aims to increase muscular explosiveness, which enables an athlete to run more quickly, leap higher, or exert force more quickly. Because it takes into account the aspects of strength, power, balance, agility, coordination, core and joint stability, foot speed, hand-eye coordination, response time, and mobility, ladder training is a multidirectional kind of exercise. During ladder training, the four fundamental abilities utilized are running, skipping, shuffling, and leaping. These ladders are lightweight and portable, making them easy to carry and use both indoors and outdoors. The player's footwork will be significantly enhanced, leading to an increase in quickness, agility, and coordination following consistent use of various speed ladder training.

DETAILED DESCRIPTION:
A team sport, cricket combines high- and low-intensity motions employing different metabolic pathways on occasion. Ladder training is a multidirectional type of exercise because it combines the elements of strength, power, balance, agility, coordination, core stability, and joint immovability. In many sports where the ability to leap, run, and change direction is required, plyometric training is used to enhance physical performance. These two have proven useful in helping athletes train for a variety of sports.

The study's goal was to compare the benefits of a plyometric training program vs a ladder training program on the agility, speed, and power of domestic female cricket players. The 42-person research sample was chosen at random. Two groups were created from the sample: group 1 received ladder training, while group 2 received plyometric training. The agility T test, the vertical leap test, and the 30-meter dash test were the result procedures. Following an 8-week course of therapy, the patients' outcome factors were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ranging from 18-25 year.
* Only female cricket players.
* Player with minimum 1- year experience of cricket.

Exclusion Criteria:

* Any cardiopulmonary problem.
* Lower extremity injuries of last 6 months(fractures, ligament ruptures).
* Players who were unable to complete ladder and plyometric training.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females of age between 18 to 25 years.
Enrollment: 42 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-07-28 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Vertical Jump test | 8 weeks
  Players stand up against a wall and use the hand that is closest to the wall to measure how high they can reach while standing. Then, using their arms and legs to propel their body higher, they do a vertical leap. The score, which is determined by subtracting their standing reach height from their jump height, is best of three attempts.
30 Yard dash test | 8 weeks
  A 30-yard sprint is required for the test, with the front foot on or behind the starting line and the shoulders parallel to the floor. Once you have held the starting stance for two seconds, you are not allowed to rock. Timing starts when the timing mechanism is triggered or the initial motion takes place.
Agility T test | 8 weeks
  The subject starts at cone A, runs to cone B, sprints there, touches the base of cone B with their right hand, shuffles sideways to cone C, then to cone D, runs back to cone B, and repeats the process until they reach cone A. The timer stops when they pass over cone A.

CONTACTS AND LOCATIONS:
Overall Officials: Sania Akram, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pechlivanos RG, Amiridis IG, Anastasiadis N, Kannas T, Sahinis C, Duchateau J, Enoka RM. Effects of plyometric training techniques on vertical jump performance of basketball players. Eur J Sport Sci. 2024 Jun;24(6):682-692. doi: 10.1002/ejsc.12097. Epub 2024 Mar 21. PMID 38874937